CLINICAL TRIAL: NCT04167397
Title: Collaboration Rather Than Isolation: Preparing Doctors of Tomorrow for Improved Medical Diagnosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Laerke Marijke Noerholk, PhD student, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: H-19063724
Record Dates: First submitted 2019-11-08; First posted 2019-11-18 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Interdisciplinary Placement
Keywords: Collaborative learning

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in permuted blocks and be allocated to either initial practice either alone or in a group of 2, 3 or 4 participants.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Single training (Experimental): Initial training individually
  Interventions: Other: Collaborative learning
- Dyad training (Experimental): Initial training in groups of 2
  Interventions: Other: Collaborative learning
- Triad training (Experimental): Initial training in groups of 3
  Interventions: Other: Collaborative learning
- Tetrad training (Experimental): Initial training in groups of 4
  Interventions: Other: Collaborative learning

INTERVENTIONS:
Other: Collaborative learning — Participants will be allocated to either single, dyad, triad or tetrad practice during initials skills training on an ultrasound simulator. Afterwards their competencies will be assessed with an individual transfer test on another simulator.

SUMMARY:
In this study, the investigators wish to explore the optimal student ratio in the simulated setting for subsequent skills transfer. The study aims to explore if there are differences in the effect of collaborative learning as a function of the number of collaborators with respect to future individual learning and transfer. Additionally, the investigators will aim to get a better understanding of the interactive processes that take place during collaborative learning. Many different theories have been used to understand collaborative learning, but few observational data have been reported in the medical literature. To gain a deeper understanding of what happens and why, the investigators plan to video record participants during their initial training and code the videos using the ICAP framework. The ICAP framework was developed by Chi in 2009 and is based on students' behaviours to reflect different modes of engagement in learning. The four behavioural modes are described as passive (P), active (A), constructive (C) and interactive (I) and each mode is associated with different examples of learning activities that can be coded. The ICAP theory proposes a hierarchical distribution of learning activities, where interactive activities are superior to constructive activities, which are superior to active activities, which are superior to passive activities (I>C>A>P). The investigators aim to investigate if this framework can serve as a conceptual framework to describe the activities that takes place during training and if these activities can be related to learning outcomes.

DETAILED DESCRIPTION:
Introduction Globally, medical schools are responding to the need for more doctors by admitting a greater number of medical students and increasing class sizes. Unfortunately, this increased intake may have detrimental effects on students' learning given the finite resources available for clinical as well as skills training. As a result, educators have called for more cost-effective methods of training and instructional methods that rely less on faculty resources than the traditional one-on-one apprenticeship model. Currently, frontline research proposes an increased focus on the role of collaborative learning in undergraduate medical education.

Recent studies have shown that collaborative learning in the form of dyad training (that is, training in pairs) compared to individual training in a simulated setting leads to improved skills transfer into the clinical workspace as well as improved skills retention. In addition, dyad training is thought to be more cost-effective than individual training because it only requires half the instructional resources, while producing similar or better educational outcomes. Concerns have been raised though, if the potentially reduced hands-on time associated with collaborative learning may affect students' learning in a negative direction over time. Therefore, examining the impact of different constellations of collaborative learning and the conditions under which the training is most effective is key to identifying when and how collaborative learning may improve students' learning outcomes.

In this study, the investigators wish to explore the optimal student ratio in the simulated setting for subsequent skills transfer. The study aims to explore if there are differences in the effect of collaborative learning as a function of the number of collaborators with respect to future individual learning and transfer. Additionally, the investigators will aim to get a better understanding of the interactive processes that take place during collaborative learning. Many different theories have been used to understand collaborative learning, but few observational data have been reported in the medical literature. To gain a deeper understanding of what happens and why, the investigators plan to video record participants during their initial training and code the videos using the ICAP framework. The ICAP framework was developed by Chi in 2009 and is based on students' behaviours to reflect different modes of engagement in learning. The four behavioural modes are described as passive (P), active (A), constructive (C) and interactive (I) and each mode is associated with different examples of learning activities that can be coded. The ICAP theory proposes a hierarchical distribution of learning activities, where interactive activities are superior to constructive activities, which are superior to active activities, which are superior to passive activities (I>C>A>P). The investigators aim to investigate if this framework can serve as a conceptual framework to describe the activities that takes place during training and if these activities can be related to learning outcomes.

Hypothesis/Research question

* Collaborative learning during initial practice leads to different levels of overt learning activities in the students. The higher level of engagement in the ICAP-hierarchy, the higher outcome on the transfer test.
* The amount of hands on time during initial practice may have effect on the immediate skills transfer

RQ: In a group of ultrasound novices, what are the effects of simulation-based obstetric ultrasound training individually, in dyads, triads or tetrads with respect to skills transfer?

Methods and Materials Study design: Controlled, randomized transfer test design Participants: Medical students will be recruited by announcements on social media (CAMES facebook page) as well as in the students' own university paper.

Inclusion criteria:

* Proficiency in the Danish language
* Passed anatomy exam of the internal genital organs
* Written informed consent

Exclusion criteria:

* Prior ultrasound experience (apart from mandatory 3 hours course in abdominal ultrasound on 6. Semester)
* Experience from gynecological/obstetric departments (work or clerkship rotation) Randomization: Randomization will be conducted using random permuted blocks. Time schedule: The project will be carried out from November 2019 and the following 8 months, with 4 months for data gathering followed by 4 months for data analysis and writing of articles.

Methods:

The participants included will be randomized to either single, dyad, triad or tetrad practice. The student(s) will start with a 10-minute video introduction to transabdominal ultrasound and biometry measurements of the fetus. Afterwards the student(s) will watch a 5-minute video introduction to the transabdominal simulator. Immediately after the student(s) will practice on a transabdominal Scantrainer (Medaphor, Ltd, Cardiff, UK), where they will train a task of assessing fetal growth during gestational ages 20-27 weeks. The training program consists of nine modules with previously established validity evidence and the measurements of Head Circumference (HC) and biparietal diameter (BPD), Abdominal Circumference (AC) and Femur Length (FL) are included in the modules. The participants will all be introduced to the simulator and the training tasks they are to complete in a similar way and will receive no further instruction during training. Technical assistance regarding the simulator will be provided if needed.

The participants will train in a fixed time frame of 2 hours, regardless of group size. They will all receive individual logins to the simulator and when training in groups they will take turn completing assignments and only one will be actively holding the ultrasound probe. Each participants' individual test scores will be saved. This training session will also be video recorded and coded according to the ICAP framework.

Immediately after completing the test the participants will undergo an individual post-test on 3 of the modules from the training session including measurements of the HC, AC and FL. The individual test scores will be saved and used for subsequent analysis and the possible identification of outliers. They will have a maximum of 15 minutes to complete this test.

Within the following week the participants will perform a transfer test on the Simbionix transabdominal simulator obtaining biometries of HC, AC and FL in a 2. trimester scanning module. Here the simulator will provide no guidance regarding optimal scanning planes and help modules. The participants will perform biometry measurements on 4 cases and the fetus will be moving during the scans as well as situated in different positions (head presentation/breach presentation). The performance will be recorded on the simulator, where the ultrasound image, the simulator buttons and the probe movements will be visible. These recordings will be scored using the OSAUS-scale (item no. 3, 4 and 5) by two expert fetal medicine experts. The participants will have maximum 10 minutes to complete each examination and the 3 measurements will be saved and compared to those of two expert fetal medicine experts, who will have completed the same scans and measurements. The use of two assessors and four cases is chosen based on a previous study demonstrating a generalizability coefficient > 0,8 with this setup.

Outcomes The primary outcome is exploring if differences in OSAUS-scores on the transfer test is related to group size during practice. The secondary outcomes is diagnostic accuracy (defined as deviation of measurements from expert ratings).

Statistics The investigators anticipate an effect size of 1,0 (Cohen's d). Using a power of 80 % and an α-value of 0,05, this corresponds to 16 participants in each study group. The investigators aim to include 20 students in each study arm to account for potential dropouts.

Publications The results are expected to be published in an international educational journal, as well as presented in medical education conferences.

Ethics Approval from the Regional Ethics Committee of the capital region of Denmark has been obtained with a letter of exemption (protocol-id: H-19063724). All participants will receive verbal as well as written information about the study and informed consent will be obtained. All participants are free to discontinue their participation at any time if the wish to do so.

ELIGIBILITY:
Inclusion Criteria:

* Proficiency in the Danish language
* Passed anatomy exam of the internal genital organs
* Written informed consent

Exclusion Criteria:

* Prior ultrasound experience (apart from mandatory 3 hours course in abdominal ultrasound on 6. Semester)
* Experience from gynecological/obstetric departments (work or clerkship rotation)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
The Objective Structured Assessment of Ultrasound Skills (OSAUS)-score | 7 days
  The primary outcome is exploring if differences in OSAUS-scores on the transfer test is related to group size during practice. The OSAUS scale consist of 7 modules and in our study the participants are only eligible to be evaluated on items no. 3, 4 and 5. Each item will be rated and generate a score between 1 and 5. This means that the participants will be able to obtain a score between 3 (minimum score) and 5 (maximum score). A high score is equivalent to a better performance than a low score.

SECONDARY OUTCOMES:
Diagnostic accuracy on biparietal diameter (BPD) | 7 days
  One of the secondary outcomes is diagnostic accuracy in measurement of BPD compared to measurements obtained by two fetal medicine experts. The measurement is in centimeter (cm).
Diagnostic accuracy on head circumference (HC) | 7 days
  One of the secondary outcomes is diagnostic accuracy in measurement of HC compared to measurements obtained by two fetal medicine experts. The measurement is in centimeter (cm).
Diagnostic accuracy on abdominal circumference (AC) | 7 days
  One of the secondary outcomes is diagnostic accuracy in measurement of AC compared to measurements obtained by two fetal medicine experts. The measurement is in centimeter (cm).
Diagnostic accuracy on femur lenght (FL) | 7 days
  One of the secondary outcomes is diagnostic accuracy in measurement of FL compared to measurements obtained by two fetal medicine experts. The measurement is in centimeter (cm).
Estimated fetal weight | 7 days
  The measurements of AC, HC and FL will be used to calculate an estimated fetal weight using the Hadlock formula:
  Weight = 10^(1,326 - (0,00326*AC*FL/100) + (0,0107*HC/10) + (0,0438*AC/10) + (0,158*FL/10). The estimated fetal weight is measured in gram (g)

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No